CLINICAL TRIAL: NCT02723214
Title: Comparison of Efficacy, Safety, Duration and Postoperative Hospitalization Between a Frameless Fiducial-less Brain Biopsy Method and the Standard Frame-based Stereotactic Biopsy
Brief Title: Comparison of Parameters Between a Frameless Brain Biopsy Method and the Standard Frame-based Stereotactic Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Miltiadis Georgiopoulos, Dr, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5807212
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Lesion of Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Frame-based stereotactic brain biopsy (Active Comparator): Brain biopsy
  Interventions: Procedure: Brain biopsy
- Frameless fiducial-less brain biopsy (Active Comparator): Brain biopsy
  Interventions: Procedure: Brain biopsy

INTERVENTIONS:
Procedure: Brain biopsy — Brain biopsy using either the frame-based stereotactic technique, or a frameless fiducial-less brain biopsy method using an optical based navigation system and a mini frame apparatus - trajectory guide.

SUMMARY:
The purpose of the present study is to compare the characteristics, i.e. efficacy, duration, safety and hospital stay, of a frameless fiducial-less brain biopsy method with those of the standard frame-based stereotactic technique.

Inclusion criteria: adult patients with cerebral lesions: 1) for whom no conclusive diagnosis could be settled in a noninvasive manner; and 2a) who also had surgically inaccessible lesions (or involving eloquent areas), or multifocal lesions, or lesions for which the probable diagnosis is a contraindication for craniotomy, or 2b) were too ill or too old for open craniotomy.

Type of Intervention: standard frame-based stereotactic brain biopsy technique or frameless fiducial-less method using an optical based navigation system and a mini frame apparatus - trajectory guide.

DETAILED DESCRIPTION:
The purpose of the present study is to compare the characteristics, i.e. efficacy, duration, safety and hospital stay, of a frameless fiducial-less brain biopsy method with those of the standard frame-based stereotactic technique, in order to apply a technique friendlier to the patient, more comfortable for the surgeon and more flexible concerning the overall hospital's function.

Inclusion criteria: adult patients with cerebral lesions: 1) for whom no conclusive diagnosis could be settled in a noninvasive manner; and 2a) who also had surgically inaccessible lesions (or involving eloquent areas), or multifocal lesions, or lesions for which the probable diagnosis is a contraindication for craniotomy, or 2b) were too ill or too old for open craniotomy.

Type of Intervention: standard frame-based stereotactic brain biopsy technique or frameless fiducial-less method using an optical based navigation system and a mini frame apparatus - trajectory guide.

The following parameters will be assessed: diagnostic yield, histological - cytological evaluation of the biopsy specimens, cerebral lesions' location, lesions' maximum diameter, duration of: the overall procedure, the preparatory steps overall, the preparation inside the OR, operation ("skin-to-skin"), the time spent inside the OR overall, neurologic morbidity, new abnormal findings in the postoperative head CT scan, length of hospitalization.

ELIGIBILITY:
Inclusion Criteria: Patients: 1) for whom no conclusive diagnosis could be settled in a noninvasive manner; and 2 who also had surgically inaccessible lesions (or involving eloquent areas), or multifocal lesions, or lesions for which the probable diagnosis is a contraindication for craniotomy.

Exclusion Criteria: 1) Pediatric patients, 2) Coagulation abnormalities, 3) destructive comorbidities and very short life expectancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic result | One month postoperatively
  Diagnostic yield, Histological - cytological evaluation of the biopsy specimens
Complications | One month postoperatively
  Neurologic morbidity, New abnormal findings in the postoperative head CT scan

SECONDARY OUTCOMES:
Length of hospitalization | One month postoperatively
Duration of the whole procedure or steps | Immediately postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Constantoyannis, MD, PhD, Study Director — Department of Neurosurgery, University Hospital of Patras, Faculty of Medicine, University of Patras

IPD SHARING:
Plan to Share IPD: No